CLINICAL TRIAL: NCT01781520
Title: Dendritic Cell/Cytokine-Induced Killer Cell Immunotherapy Combined With S-1 in Patients With Advanced Pancreatic Cancer: A Prospective Study.
Brief Title: Study of S-1 Plus DC-CIK for Patients With Unresectable Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director,Capital Medical University (CMU)Cancer Center, Capital Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1+DC CIK-P
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; S1; DC-CIK
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- S-1 plus DC-CIK (Experimental): Chemotherapy: S-1 is administered orally twice daily at a dose of 80,100, or 120mg/day for body surface areas of less than 1.25m2, between 1.25m2 and less than 1.5, or 1.5m2 or greater, respectively, for 14 consecutive days, followed by a 7-day rest, repeated every 3 weeks.
  DC-CIK Immunotherapy:Mononuclear cells were collected aseptically with blood cell separator composition aphaeresis, and then cultured DC-CIK cells were infused back to the patients on days 15, 17, and 19 of 21-day cycles.
  Interventions: Biological: DC-CIK Treatment; Drug: S1
- DC-CIK alone (Active Comparator): DC-CIK Immunotherapy:Mononuclear cells were collected aseptically with blood cell separator composition aphaeresis, and then cultured DC-CIK cells were infused back to the patients on days 15, 17, and 19 of 21-day cycles.
  Interventions: Biological: DC-CIK Treatment
- S-1 alone (Active Comparator): Chemotherapy: S-1 is administered orally twice daily at a dose of 80,100, or 120mg/day for body surface areas of less than 1.25m2, between 1.25m2 and less than 1.5, or 1.5m2 or greater, respectively, for 14 consecutive days, followed by a 7-day rest, repeated every 3 weeks.
  Interventions: Drug: S1
- Best supportive care (Active Comparator)
  Interventions: Other: Best supportive care

INTERVENTIONS:
Biological: DC-CIK Treatment — The DC-CIK cells were infused on days 15, 17, and 19 of 21-day cycles.
  Arms: DC-CIK alone; S-1 plus DC-CIK
Drug: S1 — The dose of S-1 is determined according to the body surface area as follows: <1.25 m2, 40 mg; 1.25-<1.5 m2, 50 mg; and >1.5 m2, 60 mg, given twice daily after meals for 14 days followed by a 7-day rest. Cycles is repeated every 21 days. Treatment is continued until disease progression, unacceptable toxic effects, or the withdrawal of consent.
  Arms: S-1 alone; S-1 plus DC-CIK
Other: Best supportive care — Best supportive care
  Arms: Best supportive care

SUMMARY:
The purpose of this study is to evaluate the antitumor effect and safety of clinical effectiveness S-1 plus dendritic cell activated Cytokine induced killer treatment (DC-CIK) for unresectable locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced, unresectable or metastatic adenocarcinoma of the pancreas not amenable to curative radiotherapy or surgery.
* Capable of oral intake
* Between 18 and 80 years old
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Karnofsky Performance Status (KPS) ≥ 70%
* Normal functions of heart, lung and bone marrow
* Adequate hematological profile： Hemoglobin ≥ 9.0 g/dL Absolute granulocyte count ≥ 1,500/mm3 Platelet count ≥ 100,000/mm3
* Adequate hepatic function Total bilirubin level≤ 3.0 times the upper limit of normal (ULN) Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN
* Adequate renal function(normal serum creatinine level)
* A life expectancy≥ 2 months
* Informed consent signed

Exclusion Criteria:

* Current enrollment in another clinical study with an investigational agent. Patients participating in surveys or observational studies are eligible to participate in this study
* Any radiotherapy or surgery within the previous 3 weeks
* Symptomatic brain metastasis not controlled by corticosteroids
* Bone marrow metastasis
* Active infection
* Serious complications
* Receiving a concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1: phenytoin, potassium warfarin , flucytosine, cimetidine and folinic acid.
* Pregnant or lactation women, or women with known or suspected pregnancy and men who want let to pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Treatment toxicity | 4 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v3.0

SECONDARY OUTCOMES:
The disease control rate | 4 years
  the proportion of patients who had a best response rating of complete response, partial response, or stable disease.
Progression free survival（PFS） | 4 years
  From starting date of enrollment to this study until date of first documented disease progression or date of death from any cause, whichever comes first.
Overal survival(OS) | 4 years
  From starting date of enrollment to this study until date of death from any cause
Changing trend of tumor biomarkers | 4 years
  The changing of CEA and CA-199 levels among different groups before the treatment and at the end of the first cycle of therapy
Phenotypic analysis of peripheral blood immune cells | 4 years
  Phenotypic analysis of peripheral blood mononuclear cells before the treatment and at the end of the first cycle of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Cancer Center, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Jiang N, Qiao G, Wang X, Morse MA, Gwin WR, Zhou L, Song Y, Zhao Y, Chen F, Zhou X, Huang L, Hobeika A, Yi X, Xia X, Guan Y, Song J, Ren J, Lyerly HK. Dendritic Cell/Cytokine-Induced Killer Cell Immunotherapy Combined with S-1 in Patients with Advanced Pancreatic Cancer: A Prospective Study. Clin Cancer Res. 2017 Sep 1;23(17):5066-5073. doi: 10.1158/1078-0432.CCR-17-0492. Epub 2017 Jun 13. PMID 28611200
- See also: Published article for this study — http://www.ncbi.nlm.nih.gov/pubmed/?term=Dendritic+Cell%2FCytokine-Induced+Killer+CellImmunotherapy+Combined+with+S-1+in+Patients+with+Advanced+Pancreatic+Cancer%3AA+Prospective+Study